CLINICAL TRIAL: NCT02333825
Title: Pediatric and Adolescent Patellar Instability
Acronym: PAPI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Mayo Clinic (Other); Oregon Health and Science University (Other); Inova Medical Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2014-087
Record Dates: First submitted 2014-12-12; First posted 2015-01-07 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2024-02

CONDITIONS: Patellar Instability
MeSH Terms: interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical Intervention (Other): The surgical intervention to be studied in this arm is medial patellofemoral ligament reconstruction surgery using hamstring tendon. The tendon used will generally consist of autograft semitendinosus. If the hamstrings have been previously harvested or injured (i.e. in the setting of anterior cruciate ligament reconstruction or proximal tibial surgery), or if the patient/his or her family prefers to minimize donor site morbidity, allograft may be used.
  Interventions: Procedure: Medial patellofemoral ligament reconstruction surgery
- Conservative treatment (Other): The intervention to be studied in this arm is a rehabilitation program directed by physical therapists. If patients in this arm are found to have a small loose body, a simple arthroscopy will be performed to remove the loose body, but no stabilization of the patellofemoral joint will be performed. The rehabilitation program will be compiled into a booklet and distributed for use by the physical therapist chosen by the patient.
  Interventions: Other: Physical therapy and rehabilitation

INTERVENTIONS:
Procedure: Medial patellofemoral ligament reconstruction surgery — Medial patellofemoral ligament reconstruction surgery using hamstring autograft
  Other Names: CPT code: 27427
  Arms: Surgical Intervention
Other: Physical therapy and rehabilitation — A standardized physical therapy and rehabilitation program to be administered and guided by rehab specialists
  Arms: Conservative treatment

SUMMARY:
This is a multi-center, randomized controlled clinical trial, the purpose of which is to determine if patients age 25 and younger who undergo medial patellofemoral ligament (MPFL) reconstruction have lower rates of recurrent instability compared to those treated non-operatively. The MPFL is a ligament that stabilizes the kneecap, and maintains its proper position in the groove on the femur (thighbone). Instability refers to a situation in which the kneecap moves out of place, or dislocates. When instability is recurrent, it occurs more than once in the same knee.

DETAILED DESCRIPTION:
A total of 240 patients will be enrolled across participating sites around the country. These sites currently include: The Hospital for Special Surgery, Oregon Health and Science University, Inova Sports Medicine, and Mayo Clinic. Patients are randomly assigned to one of two treatment groups. Patients assigned to the "stabilization" group will undergo surgery to reconstruct the MPFL using either a hamstring tendon that is your own or one obtained from a donor. Patients assigned to the "conservative" group will be treated with physical therapy, and possibly a simple knee arthroscopy if you are found to have a loose fragment on x-ray or MRI. All patients will be required to return for follow-up visits, which will continue over the course of 5 years. During these visits, patients will be examined, asked to answer questions about their surgery and general health, and have imaging (x-ray and MRI) performed on the knee. All patients enrolled in this study will undergo a standardized, intensive rehabilitation protocol. The investigators anticipate that all patients may benefit from extensive rehabilitation, including strengthening and return to sport training. The knowledge gained from this study may benefit others in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be age 25 or younger
* Patients must be first-time dislocators, meaning have had only one episode of patellar instability, during which they dislocated their patella (kneecap)

Exclusion Criteria:

* Patients with more than one episode of patellofemoral instability
* Patients who have had prior patellofemoral surgery on the knee of interest
* Patients with large cartilage tears in the knee. These patients will undergo stabilization of the patellofemoral joint (MPFL reconstruction) as per standard of care, and will not be included in the study.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of patellar instability | 5 years
  The primary outcome is recurrent episode of patellar instability within 5 years following the primary patellofemoral dislocation event. A preliminary analysis will be performed at 2 years to examine for any early results of the study. Patellar instability will be defined as any patient-reported episode of subluxation or dislocation following the index event. Subluxation or dislocation will be defined as a feeling of dissociation of the patella from its trochlear groove. Subluxation will be noted if the patella spontaneously reduces into the groove, and dislocation will be noted if the patella requires any change in position or force (i.e. extending the knee or exerting a medially-directed force on the patella) in order to reduce into its trochlear groove. (Apprehension will not be classified as subluxation unless the patient specifically notes a sensation of departure of the patella from its trochlear groove at some point during the experience.)

SECONDARY OUTCOMES:
Kujala Scoring Questionnaire | Preoperatively and at 1 year, 2 years, 3 years, 4 years, and 5 years after treatment.
  The Kujala Scoring Questionnaire is a validated patient reported outcome measure
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Preoperatively and at 1 year, 2 years, 3 years, 4 years, and 5 years after treatment.
  The KOOS is a validated patient reported outcome measure
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation | Preoperatively and at 1 year, 2 years, 3 years, 4 years, and 5 years after treatment.
  The IKDC Subjective Knee Evaluation is a validated patient reported outcome measure
Hospital for Special Surgery Pediatric Functional Activity Brief Scale | Preoperatively and at 1 year, 2 years, 3 years, 4 years, and 5 years after treatment.
  The Hospital for Special Surgery Pediatric Functional Activity Brief Scale is a validated patient reported outcome measure
Outerbridge grade of any cartilage lesions | MRI taken at initial exam, and for patients randomized to surgery only at 1 year and 5 years after surgery as well
  Outerbridge grade will be used to describe the severity of articular cartilage lesions at initial presentation and for surgical patients, 1 and 5 years after treatment as well

CONTACTS AND LOCATIONS:
Overall Officials: Beth E Shubin Stein, MD, Principal Investigator — Hospital for Special Surgery, New York; Jacqueline Munch, MD, Study Chair — Oregon Health and Science University Hospital; Diane Dahm, MD, Study Chair — Mayo Clinic; Robin V West, MD, Study Chair — Inova Sports Medicine

REFERENCES:
- See also: Principle Investigator: Beth Shubin Stein, MD — http://www.hss.edu/physicians_shubin-stein-beth.asp